CLINICAL TRIAL: NCT01090089
Title: The Combination of Lenalidomide and Dexamethasone With or Without Intensification by High-dose Melphalan in the Treatment of Multiple Myeloma
Brief Title: Combination of Lenalidomide and Dexamethasone in Treatment of Multiple Myeloma
Acronym: DSM XIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSMM XIII
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenalidomid, PBSCT (Experimental): A1 Rd until progression or max. 5 years (Rd = lenalidomide 25 mg d1-21/28d + dexamethasone 40 mg po d1, d8, d15, d22/28d)
  Interventions: Drug: Lenalidomide, Dexamethasone, PBSCT
- Lenalidomid (Active Comparator): A2 Induction with 3 cycles Rd, tandem high dose melphalan (140 mg/m²) with autologous peripheral blood stem cell transplantation (PBSCT) followed by lenalidomide maintenance (10 mg/day) until progression or max. 5 years
  Interventions: Drug: Lenalidomide, Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide, Dexamethasone — Rd until progression or max. 5 years (Rd = lenalidomide 25 mg d1-21/28d + dexamethasone 40 mg po d1, d8, d15, d22/28d)
  Other Names: Revlimid
  Arms: Lenalidomid
Drug: Lenalidomide, Dexamethasone, PBSCT — Induction with 3 cycles Rd, tandem high dose melphalan (140 mg/m²) with autologous peripheral blood stem cell transplantation (PBSCT) followed by lenalidomide maintenance (10 mg/day) until progression or max. 5 years
  Other Names: Revlimid
  Arms: Lenalidomid, PBSCT

SUMMARY:
In this study for elderly myeloma patients lenalidomide plus low-dose dexamethasone until progression is being compared with age-adjusted tandem high-dose melphalan 140 mg/m² augmented by induction with 3 cycles of lenalidomide plus low-dose dexamethasone before transplantation and lenalidomide maintenance after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form. 2. Age 60-75 years at the time of signing the informed consent form. 3. Able to adhere to the study visit schedule and other protocol requirements. 4. Symptomatic MM requiring therapy. 5. Measurable monoclonal protein in serum and/or urine 6. Monoclonal plasma cells in the bone marrow >/= 10% and/or biopsy-proven plasmacytoma 7. Myeloma-related organ dysfunction, at least one of [C] Calcium elevation in the serum (> 11.5 mg/dL or > 2.65 mmol/l) [R] Renal insufficiency (creatinine > 173 μmol/l or > 2 mg/dL) [A] Anemia (Hb < 10 g/dL or 2 g/dL < normal) [B] Bone lesions or general osteoporosis 8. ECOG PS of </= 2 ... 9. Laboratory test results within these ranges within 1 week prior to randomization:

* ANC >/= 1.0 x 109/L.
* Platelet count >/= 75 x 109/L or in case of bone marrow infiltration with myeloma cells >/= 30 x 109/L.
* Total bilirubin </= 2 mg/dL.
* AST (SGOT) and ALT (SGPT) </= 3 x ULN. 8. Female subjects of childbearing potential must: o Understand the study drug is expected to have a teratogenic risk

  o Agree to use, ..., effective contraception without interruption,...

  o Understand that even if she has amenorrhea, she must follow all the advice on effective contraception.

  o She understands the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy

  o Agree to have a medically supervised pregnancy test ...
* Male subjects must

  o Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study drug therapy ...
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* All subjects must

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study drug with another person and to return all unused study drug to the investigator.

    9. Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.

    10. Able to receive antithrombotic prophylaxis (...). 11. Life-expectancy > 3 months.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the ICF.
2. Pregnant or lactating females
3. Any condition, incl. the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Patient currently is enrolled in another clinical research study or has been enrolled ...within 4 weeks before randomization and/or is receiving an investigational agent for any reason ...
5. Known hypersensitivity to thalidomide, dexamethasone, or melphalan.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or active infectious hepatitis, type A, B or C or treponema pallidum
10. Prior treatment with dexamethasone discontinued because of ≥ grade 3 dexamethasone-related toxicity.
11. Any prior chemotherapy with the exception of a short course of dexamethasone more than 4 weeks before randomization.
12. Immunotherapy or antibody therapy within 8 weeks before randomization.
13. Major surgery within 4 weeks before randomization.
14. Renal failure requiring dialysis.
15. Myocardial infarction within 6 months before randomization, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
16. Severe pulmonary disease (diffusion capacity < 60% of normal).
17. Treatment for cancer other than MM within 5 years before randomization, with the exception of basal cell carcinoma or cervical cancer in situ.
18. Cardiac amyloidosis.
19. Poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to the protocol.
20. Any systemic infection requiring treatment.
21. Unability or unwillingness of the patient to receive antithrombotic prophylaxis.

    -

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 yrs
  To compare the efficacy of both treatment regimens with regard to progression-free survival.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 yrs
  To assess the safety and overall survival of both treatment regimens.
• Response (complete response [CR], stringent complete response [sCR], very good partial response [VGPR], partial response [PR] and overall response [CR (incl. sCR)+ VGPR + PR]) according to IMWG criteria | 5 yrs
  To investigate other efficacy parameters of both treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Christian Straka, Principal Investigator — Agirov Klinik
Locations (31):
- Germany (31):
  - Universitätsklinikum Münster, Münster, North Rhein Westfallen
  - Universitätsklinikum Aachen, Aachen
  - Agirov Klinik, Berg
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Klinikum Bremen-Mitte, Bremen
  - Universitätsklinik Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität Greifswald -Anstalt öffentlichen Rechts-, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Stiftungsklinikum Mittelrhein gGmbH, Koblenz
  - Klinikum Landshut gemeinnützige GmbH, Landshut
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Hämato-Onkologische Schwerpunktpraxis, München
  - Onkologische Praxis Elisenhof, München
  - Klinikum München Harlaching, München
  - Klinikum rechts der Isar, München
  - Klinikum Nord, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie und Onkologie, Ravensburg
  - Klinikum der Universität Regensburg, Regensburg
  - Diakonie-Klinikum Stuttgart-Diakonissenkrankenhaus und Paulinenhilfe gGmbH, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Universitätsklinikum Ulm, Ulm
  - HSK Dr. Horst-Schmidt-Kliniken gmbh, Wiesbaden
  - Universitätsklinikum Würzburg, Würzburg